CLINICAL TRIAL: NCT00983099
Title: Evaluation of Pharmacokinetics, Safety and Tolerability of Single and Multiple Oral Doses of Neramexane Mesylate in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Manager Public Disclosure, Merz Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MRZ 92579/NA/1006
Record Dates: First submitted 2009-09-18; First posted 2009-09-23 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
MeSH Terms: interventions — neramexane

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Neramexane — single and multiple dose, tablets, oral

SUMMARY:
Part 1 (single dose)

Primary parameters

* Area under the plasma concentration curve from zero to infinity [AUC0-inf] and observed maximum plasma concentration [Cmax] of Japanese and Caucasian subjects for each dose group
* If at least 20% of the Japanese or of the Caucasian subjects have an area under the plasma concentration curve extrapolation [AUCextrap%] >20% relative to AUC0-inf for one of the dose groups area under the plasma concentration curve from zero to the last measurable concentration [AUC0- tz] becomes primary parameter for Japanese and Caucasian subjects for all of the dose groups. In this case AUC0-tau will become a secondary parameter

Secondary parameters and derived values from statistical analysis

* Dose proportionality and linearity in Japanese subjects
* Ratios (Japanese vs. Caucasian subjects) of AUC0-∞ and Cmax for each dose group
* Dose normalized AUC [AUC0-inf,norm], dose normalized Cmax [Cmax,norm], AUC0- tz, time of occurrence of Cmax [tmax], apparent terminal half life [t½], mean residence time [MRT], apparent (oral) total plasma clearance [CLtot/f], apparent volume of distribution during the terminal disposition phase [Vz/f], AUCextrap%, apparent terminal disposition rate constant [λz], weight corrected AUC0-inf, weight corrected AUC0-tz, weight corrected Cmax, weight corrected CLtot/f, cumulative amount of excreted Neramexane into urine [Ae0-tz], fraction of orally administrated drug excreted into urine [fe/f], renal clearance [CLR] and apparent non-renal clearance [CLNR/f]
* Safety and tolerability

Other parameters

* Pharmacogenetics
* Amount of N-OH Neramexane excreted in urine [Ae0-tz] if a validated method will be available at the time of analysis
* Metabolite determination (N-OH Neramexane) in plasma and urine, optional (may be analyzed and evaluated if a validated method will be available at the time of analysis)
* Endogenous creatinine clearance [CLCR], amount of excreted creatinine into urine per hour [AeCR,hr]
* Evaluation of further metabolites will be described in detail in the Statistical Analysis Plan

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* Caucasian (Part 1 only) or Japanese origin
* Japanese subjects must have a Japanese passport, Japanese grandparents and parents and not have lived outside of Japan for more than 5 years
* Aged 20 to 55 years (inclusive)
* Body weight between 50 and 90 kg (inclusive) with BMI ranging from 18.0 to 28.0 kg/m2 (inclusive) Japanese females may have a body weight of at least 45 kg (inclusive) with BMI ranging from 17.0 to 28.0 kg/m2 (inclusive)
* Females must have a negative urine pregnancy test at screening and on Day -1 for Part 1 and on Day 1 for Part 2
* Subjects must be willing to use one of the following methods of contraception from the first dose of trial medication until completion of follow-up procedures.

  * All subjects must agree to use condom and spermicide.
  * Male subjects without vasectomy (with documentation of azoospermia) must assure that their female partners uses another form of contraception such as non hormonal IUD, diaphragm.
  * Female subjects of childbearing potential must agree to use an effective method of birth control such as sexual abstinence, vasectomised partner, non hormonal IUDs or double contraception methods (e.g., condom with spermicide cream) from Screening until one month after last application of study drug.
* Willing and able to give written informed consent after having been informed of the requirements and the restrictions of the study

Exclusion Criteria:

* Subjects who have taken part in the drug administration phase of the single dose part are excluded from participation in the multiple dose part of the study and vice versa
* Any clinically relevant finding on medical history or, physical examination affecting subject's safety or the study objectives
* Any disease or condition, which could influence the physiological absorption, distribution and metabolic turnover (e.g. endocrine diseases, febrile conditions, severe infections, acute inflammations, chronic diarrhoea, chronic vomiting, gastrointestinal disease or surgery of the gastrointestinal tract, including cholecystectomy); appendectomy older than 6 months is allowed
* Prior history or present evidence of clinically significant metabolic, renal, hepatic, pulmonary or cardiovascular disease, CNS disorders or disturbances of bleeding (hemorrhagic diathesis), diagnosis of malignancy, polyneuropathy or psychiatric disorder, organ transplantation
* Any clinically relevant abnormal laboratory value (haematology, clinical chemistry, urinalysis) or laboratory values which in the discretion of the investigator and the Merz scientific expert might affect subject's safety or the study objectives
* Positive serology for human immunodeficiency virus [HIV] (HIV1/HIV2 antibodies), hepatitis B surface antigen [HBsAg], antibodies against hepatitis C virus [anti-HCV]
* Clinically relevant abnormalities in the 12-lead ECG which in the discretion of the investigator and the Merz scientific expert might affect the study objectives
* Presence or history of clinically relevant allergy or a known or suspected hypersensitivity to Neramexane, Memantine or Amantadine and/or its study medication excipients and to quinine hydrochloride (slight seasonal hay fever is allowed as long as the season does not meet the study period)
* History of alcohol or drug dependence
* Alcohol consumption averaging more than 40 g alcohol (4 units) daily (28 units per week) within the last year for males and more than 20 g (2 units) daily within the last year for females
* Regular caffeine consumption averaging more than 5 cups of coffee or equivalent (500mg caffeine) per day within the last year
* Smoking more than 5 cigarettes per day or equivalent (use of snuff, nicotine replacement chewing tobacco)
* Refusal or inability to eat the meals provided by the clinic (e.g. vegetarian)
* Nursing mother
* Woman planning pregnancy during the course of the trial
* Evidence or suspicion that the subject might not comply with the study directives and/or that he/she is not reliable or trustworthy
* Evidence or suspicion that the subject is not willing or unable to understand the information that is given to him/her as part of the informed consent, in particular regarding the risks and discomfort to which he/she would agree to be exposed
* Subjects who are imprisoned or are lawfully kept in an institution
* Employees or direct relatives of an employee of the CRO or Merz Pharmaceuticals
* Systolic blood pressure <90 mm Hg or >140 mm Hg or diastolic blood pressure <50 mm Hg or > 95 mm Hg in supine position
* Pulse rate < 45 or > 100 beats per minute [bpm]
* Use of any prescribed drugs in the 4 weeks prior to the first administration of the IMP
* Regular use of over-the-counter [OTC] drugs (except paracetamol, maximum 1 g/day) in the 4 weeks prior to the first administration of the IMP or at least 10 half lives, whichever is longer
* Occasional use of OTC drugs (except paracetamol, maximum 1 g/day) in the 2 weeks prior to the (first) administration of the IMP
* Females taking hormonal contraceptives
* Participation in another clinical study of any IMP within 2 months prior to the first administration of IMP
* History of blood loss or donation of blood or plasma exceeding 450 ml within the last 3 months before first administration of IMP
* Acute illness in the past 14 days before administration of IMP (Day 1)
* Fever (oral > 37.5 °Celsius or 99.5 °Fahrenheit, respectively) in the last 8 days before Day 1 as reported by history or on Day 1
* Alcohol intake within the last 48 hours prior to the (first) administration of the IMP and a positive alcohol breath test on Screening and Day-1 for Part 1 and on Day 1 for Part 2
* Intake of recreational drugs within the last 4 weeks prior to first administration of IMP on Day 1 and a positive urine test for drugs of abuse on screening, Day -1 for Part 1 and Day 1 for Part 2
* Consumption of xanthine containing food or beverages within the last 48 hours prior to the first administration of the IMP
* Consumption of herbs/fruits that can have an influence on pharmacokinetics such as St. Johns wort, grapefruits or grapefruit juice within the last 72 hours prior to the first administration of the IMP

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determination of plasma concentration after single and multiple dose | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- California Clinical Trials, Glendale, California, United States